CLINICAL TRIAL: NCT06530979
Title: The Effectiveness of a Tailored Nutritional Education Program Utilizing Saudi-Sign Language on Adults With Profound Hearing Impairment
Brief Title: The Effectiveness of a Tailored Nutritional Education Program on Profound Hearing Impairment Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Jenan Aljubair, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: kingSaudU1
Record Dates: First submitted 2024-07-08; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Profound Hearing Impairment; Nutrition, Healthy
Keywords: Profound hearing impairment; Nutrition knowledge; Nutrition status; Intervention nutrition education

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional education program intervention (Experimental): Nutritional education program intervention (NEP group n=30) profound hearing-impaired people who will receive tailored nutritional education program intervention utilizing Saudi-Sign Language supplied by a sign language interpreter in the videos and person during sessions.
  Interventions: Device: Tailored nutritional education program utilizing Saudi-sign language supplied by Saudi-sign language interpreter
- Control (No Intervention): Control (C group n=31) Profound hearing-impaired people who will non- receive tailored nutritional education program intervention utilizing Saudi-Sign Language

INTERVENTIONS:
Device: Tailored nutritional education program utilizing Saudi-sign language supplied by Saudi-sign language interpreter — The program will be implemented in an experimental group composed of profoundly impaired hearing adults (91 Decibels and above). The experimental group will receive nutrition group counselling via photos, and models, and Saudi-sign language interpreter, including awareness of food groups and their nutrients, choose healthy and balanced items from supermarkets, restaurants or coffee shop menus-traffic lights on nutrition labelling and health problems or diseases related to diet and weight management
  Arms: Nutritional education program intervention

SUMMARY:
Literature suggests that profound hearing-impaired people have poor access to health care directly related to communication difficulties. A lack of knowledge regarding health and healthy dietary patterns has been documented. Several associations between chronic diseases such as obesity, CVD, hyperlipidemia etc., and hearing impairments have been established. There is a gap in the literature for studies that use Saudi-sign language-tailored programs in patient health and nutrition education.

This project aims to create a Saudi-sign language general nutritional education program and then test its effectiveness in enhancing the nutritional status and knowledge of Saudis with profound hearing impairments.

DETAILED DESCRIPTION:
Literature suggests that profound hearing-impaired people have poor access to health care directly related to communication difficulties. A lack of knowledge regarding health and healthy dietary patterns has been documented. Several associations between chronic diseases such as obesity, CVD, hyperlipidemia etc., and hearing impairments have been established. There is a gap in the literature for studies that use Saudi-sign language-tailored programs in patient health and nutrition education.

This project aims to create a Saudi-sign language general nutritional education program and then test its effectiveness in enhancing the nutritional status and knowledge of Saudis with profound hearing impairments.

Methods: The study will be divided into two phases. The first phase will cultural adaptation and translation of the General Nutrition Knowledge Questionnaire (GNKQ) which will be used in the intervention study. In this phase, the forward-backwards technique will be followed, for internal consistency will be used Cronbach's alpha. A Saudi-sign language general nutritional education program will be created from accredible source for content appropriateness. For the second phase, the interventional study, the participants will be randomly selected and allocated to either the control or the experimental group. The efficacy of the Saudi-sign language general nutrition education program to enhance the knowledge and nutrition health of Saudi adults with profound hearing impairment will be compared to a control group. A small group counselling will be delivered to the experimental group using pictures, animated films, models, and Saudi-sign language translations supplied by a sign language interpreter in the videos and person during sessions. The same video will be used to create PowerPoint with nutritional education information for the control group in Arabic. Anthropometric data, body composition, a 3-day food diary, and the GNKQ will all be gathered at baseline and twelve weeks later.

ELIGIBILITY:
Inclusion Criteria:

1. Saudi adults
2. Aged between 18-65 years
3. Both males and females
4. Known case of profound hearing impairment /disability
5. knowledgeable in Saudi Sign Language.

Exclusion Criteria:

1. Aged <18 years
2. Not knowing the Saudi Sign Language
3. Other disabilities such as mental or physical disability
4. Have nutritional knowledge such as attended course/s related nutrition or studied in nutrition field
5. Illiterate
6. Pregnant or planning a pregnancy, or on breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-03-02 (Estimated)

PRIMARY OUTCOMES:
Nutrition knowledge | 3 months
  General Nutrition Knowlege Questionnaire GNKQ as videos used Saudi Sign language (Multiple-choice questions with a single select multiple choice question).
Anthropometric measurements | 3 months
  Anthropometric measurements (e.g., weight and height will be combined to report BMI in kg/m^2), (Wist and hip circumference will be combined to report Wist/Hip ratio).
Body composition measurement | 3 months
  Body composition measurement via Tanita to measure (FM, FFM, Muscle mass in Kg and TBW %).
Dietary assessment | 3 months
  A 3-day food record diary (two days weekday and one day weekend).

CONTACTS AND LOCATIONS:
Overall Officials: Jenan Aljubair, Ph.D, Principal Investigator — King Saud University
Locations (1):
- College of Applied Medical Sciences, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No